CLINICAL TRIAL: NCT06873581
Title: A Pivotal Study of Voro Urologic Scaffold for the Treatment of Post Prostatectomy Stress Urinary Incontinence (ARID II)
Brief Title: Pivotal Study of Voro Urologic Scaffold
Acronym: ARID II
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Levee Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1010174
Record Dates: First submitted 2025-03-07; First posted 2025-03-12 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Radical Prostatectomy; Stress Urinary Incontinence (SUI)
Keywords: SUI; Radical Prostatectomy; Voro Urologic Scaffold; ARID II; Post-prostatectomy incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Intervention Model Description: This is a multicenter, single blind, randomized controlled study.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Voro Urologic Scaffold Group (Experimental): Participants will undergo robotic assisted radical prostatectomy procedure as part of their standard of care treatment for their prostate cancer. The Voro Urologic Scaffold will be placed during the prostatectomy procedure after prostate removal.
  Interventions: Device: Voro Urologic Scaffold
- Control Group (No Intervention): Participants will undergo robotic assisted radical prostatectomy procedure as part of their standard of care treatment for their prostate cancer. This group will not receive Voro Urologic Scaffold during the treatment.

INTERVENTIONS:
Device: Voro Urologic Scaffold — The Voro Urologic Scaffold is placed during the prostatectomy procedure after prostate removal.
  Arms: Voro Urologic Scaffold Group

SUMMARY:
The objective of this study is to compare safety and effectiveness of the Voro Urologic Scaffold in adult men undergoing robotic assisted radical prostatectomy as compared to control arm.

The study is a multi-center, single blind, randomized, controlled trial. Up to 266 participants will be treated at up to 30 centers in the United States. The study will consist of a Baseline visit, implantation during robotic assisted radical prostatectomy (RARP), catheter removal, 6 weeks, 6 months, 12 months, 18 months, and 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Male >= 45 years of age of any race and ethnic group
2. Diagnosed with prostate cancer and scheduled for radical prostatectomy
3. Gleason Grade Group 4 or lower
4. Prostate size less than 80 grams, as measured by Magnetic Resonance Imaging (MRI)
5. Able and willing to provide written consent to participate in the study
6. Able and willing to comply with study follow-up visits and procedures
7. Willing to forego any other procedures for stress urinary incontinence (SUI) during the study

Exclusion Criteria:

1. Malignant tumors with known bladder neck or urethral sphincter invasion or metastatic disease confirmed via baseline assessments (example [e.g.,] Multiparametric magnetic resonance imaging [mpMRI], bone scan)
2. History of urinary incontinence, including stress or urge urinary incontinence
3. Demonstration of SUI, such as positive 1 hour pad weight test or participant reported incontinence episodes
4. Currently treated with medications to treat overactive bladder (OAB)
5. Post void residual >200 milliliter (ml) or > 25 percentage (%) total volume(= voided volume + residual volume)
6. Presence of urethral stricture or bladder neck contracture
7. History of urethral stricture
8. Current or chronic urinary tract infection
9. Prior urologic outlet surgical or minimally invasive procedure (e.g., Transurethral resection of the prostate [TURP], Holmium laser enucleation of the prostate [HoLEP,] Rezum, etc.).
10. Prior pelvic radiation or anticipated need for radiation after radical prostatectomy
11. History of neurogenic lower urinary tract dysfunction
12. History or current need for intermittent urinary catheterization
13. Body mass index >40
14. History of cancer (excluding prostate cancer meeting the inclusion criteria) which is not considered in complete 5 year remission (excluding squamous and basal cell skin carcinoma)
15. History of bladder malignancy
16. Diagnosed or suspected primary neurologic conditions known to affect voiding function
17. History of clinically significant congestive heart failure (i.e., New York Heart Association [NYHA] Class III and IV)
18. Current uncontrolled diabetes (i.e., hemoglobin A1c [glycated hemoglobin or glycosylated hemoglobin] >=7.5%)
19. Current overactive bladder defined as a score of > 8 on the Overactive Bladder Questionnaire (OAB-8) administered at the baseline visit
20. History of immunosuppressive conditions or on medications which modulate the immune system
21. Any significant medical history that would pose an unreasonable risk or make the participant unsuitable for the study per investigator discretion
22. Participant with planned concomitant surgery
23. Anterior fascial sparing radical prostatectomy
24. Retzius sparing radical prostatectomy
25. Participant currently participating in other investigational studies unless approved by the Sponsor in writing
26. Participant is, in the investigator's judgement, part of a vulnerable population, including but not limited to:

    1. Prisoners
    2. Individuals pending incarceration
    3. Individuals experiencing any cognitive or psychiatric condition that interferes with or precludes direct and accurate communication with the study investigator regarding the study or affects the ability to complete the study quality of life questionnaires
27. Planned adjuvant radiation therapy

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 266 (Estimated)
Dates: Start 2025-04-18 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | Upto 24 months
  AE is any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in participants during the course of the study, whether or not related to the investigational device.
Number of Participants With Adverse Events Categorized by Severity | Upto 24 months
  The severity of adverse events as assessed by the investigator; events will be based on the definitions outlined in the Common Terminology Criteria for Adverse Events (CTCAE) v5.0.
Number of participants achieving continence as measured by 1 hour provocative pad weight test at 6 weeks post-prostatectomy | At 6 weeks post-prostatectomy

SECONDARY OUTCOMES:
Severity of incontinence as measured by 1 hour provocative pad weight test at 6 weeks | At 6 weeks
Severity of incontinence as measured by 1 hour provocative pad weight test at 6 months | At 6 months
Quality of Life (QoL) performance as assessed by the urinary domain of Expanded Prostate Cancer Index Composite (EPIC) Questionnaire | At 6 weeks, 6 months and 12 months
  The Expanded Prostate Cancer Index Composite is a validated, comprehensive questionnaire designed to evaluate patient function and bother after localized prostate cancer treatment. Response options for each item form a Likert scale, and multi-item scale scores are transformed linearly to a 0-100 scale, with higher scores representing better quality of life.
Continence rate as measured by 1-hour provocative pad weight test at 6 months post-prostatectomy | At 6 months post-prostatectomy
Number of participants achieving continence as measured by 1 hour provocative pad weight test at 12 months post-prostatectomy | At 12 months post-prostatectomy

CONTACTS AND LOCATIONS:
Overall Officials: Karen Cornett, Study Director — Vice President, Levee Medical, Inc
Locations (20):
- United States (20):
  - Mayo Clinic, Phoenix, Arizona
  - Academic Urology, Sun City, Arizona
  - UCLA Urology, Los Angeles, California
  - University of California San Diego, San Diego, California
  - Tampa General Hospital, Tampa, Florida
  - University of Chicago Medicine, Chicago, Illinois
  - IU school of Medicine, Department of Urology, Indianapolis, Indiana
  - University of Maryland, Baltimore, Maryland
  - John Hopkins, Baltimore, Maryland
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - BMHCC/ Mississippi Urology Clinic, Jackson, Mississippi
  - Northwell Health, New Hyde Park, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Erlanger Urology, Chattanooga, Tennessee
  - The Conrad Pearson Clinic, Germantown, Tennessee
  - Urology Associates PC Nashville, Nashville, Tennessee
  - Urology of Austin, Austin, Texas
  - Potomac Urology Center, Alexandria, Virginia
  - Urology of Virginia, PLLC, Virginia Beach, Virginia

IPD SHARING:
Plan to Share IPD: No